CLINICAL TRIAL: NCT00295412
Title: The Impact of Quetiapine on the Drug Abuse Patterns of Addicted Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5077-99904
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2006-02-23 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Substance Use Disorders
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders | interventions — Quetiapine Fumarate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: quetiapine (drug)

SUMMARY:
The lifetime of substance use disorders in schizophrenia is close to 50%. Substance abuse in schizophrenia is associated with negative consequences. Unfortunately, there no clear guidelines for the pharmacological treatment of this dual diagnosis population. Preliminary results suggest that second-generation antipsychotic drugs (mainly clozapine) may relieve drug cravings in schizophrenia. We performed a 12-week pilot study to evaluate the impact of quetiapine, a second-generation antipsychotic, on substance abuse parameters, psychiatric symptoms and side effects in patients schizophrenia and comorbid substance use disorders. Our expectation was a 20 % decrease in drug cravings from baseline to end-point.

ELIGIBILITY:
Inclusion Criteria:

* Patients with as schizophrenia spectrum disorder
* Patients with a comorbid substance use disorder

Exclusion Criteria:

* Patients already on quetiapine or clozapine
* Patients hospitalized or acutely ill
* Total score lower than 65 on the PANSS
* Pregnancy
* Female subjects of childbearing potential without adequate contraception
* Abnormal liver function (hepatic enzymes more than 3 times the upper normal limits)
* Any clinically meaningful unstable renal, hepatic, cardiovascular, respiratory, cerebrovascular disease or other serious, progressive physical disease.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Stip, Md, MSc, CSPQ, Principal Investigator — Centre de recherche Fernand-Seguin, Hôpital Louis-H Lafontaine, Departement of Psychiatry, Faculty of medicine, University of Montreal
Locations (1):
- Centre de recherche Fernand-Seguin, Montreal, Quebec, Canada